#### HONG KONG METROPOLITAN UNIVERSITY

#### **Information Sheet**

#### TITLE OF THE STUDY

Effect of inspiratory muscle training on respiratory function, diaphragm thickness, balance control, exercise capacity and quality of life in people after stroke: a randomized controlled trial

#### INTRODUCTORY SENTENCE

You are invited to participate in a research study conducted by Prof. William Tsang Wai Nam from the Department of Physiotherapy, School of Nursing and Health Studies of Hong Kong Metropolitan University (HKMU).

#### **PURPOSE OF THE STUDY**

(1) Based on the optimal inspiratory muscle training (IMT) intensity identified from our previous study, this randomized controlled trial (RCT), aims to explore the effects of different training surfaces during a 4-week IMT protocol on inspiratory function, balance control, exercise capacity, and quality of life in people after stroke (2) To ascertain the effect of IMT on the relationship between diaphragm muscle contraction and activation of other trunk muscles.

#### **PROCEDURES**

In this study, you will be randomly allocated into three groups to receive IMT with different intensity. Apart from IMT, all groups will also receive the same conventional rehabilitation. All interventions will be implemented 5 days per week for 4 weeks. We will assess your respiratory function, diaphragmatic function, balance control, walking capacity, QOL and trunk muscle activity before and after 4 weeks intervention. After 12 weeks follow-up after the end of intervention partial outcomes will be measured again.

All measurements and training in this study are non-invasive.

# POTENTIAL RISKS/STRESS/PAIN/DISCOMFORTS/OTHER FACTORS AND THEIR MINIMIZATION

There will be no direct risk, stress, pain or discomforts in participating in this study.

#### POTENTIAL BENEFITS

There will be no direct benefit in participating in this study.

#### PARTICIPATION AND WITHDRAWAL

You have every right to withdrawn from the study before or during the measurement without

penalty of any kind.

#### **CONFIDENTIALITY**

Your personal information and data will not be disclosed to any person not being in the research team. Your name or photo will not appear on any published materials.

#### **QUESTIONS AND CONCERNS**

If you have any questions or concerns about the research study, please feel free to contact Prof William Tsang Wai Nam of HKMU at 3970 8703. If you have questions about your rights as a participant of this research study, please contact the Research Ethics Committee of HKMU at 2768 6251.

# **Consent Form**

## Hong Kong Metropolitan University School of Nursing and Health Studies, Department of Physiotherapy

### Consent form for

| Effect of inspiratory muscle training on respiratory function, diaphragm thickness, balance |
|---|
| control, exercise capacity and quality of life in people after stroke: a randomized controlled |
| trial |

| trial I have read and understand the information provided about the above study. I agree to participate to this study. | |
|---|---|
| Name of investigator | Signature of investigator |